CLINICAL TRIAL: NCT06668363
Title: Enhancing HIV Prevention and Reducing Alcohol Use Among People Receiving STI Care in Lilongwe, Malawi: A Pilot Implementation Study
Brief Title: Enhancing HIV Prevention and Reducing Alcohol Use Among People Receiving STI Care in Lilongwe, Malawi
Acronym: Treat4All
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24-1648; R34AA030939 (NIH)
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Alcohol Consumption; PrEP Uptake; Recent Heavy Drinking; HIV Prevention; HIV Treatment
Keywords: PrEP; HIV; HIV Prevention; Alcohol reduction; Alcohol
MeSH Terms: conditions — Alcohol Drinking | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Data analysts will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treat4All (Experimental): Treat4All will be based on Fleming's Project TrEAT, culturally adapted to the Malawi context, and enhanced to include content on HIV prevention and treatment activities (PrEP use for those at risk for HIV; ART adherence and viral suppression for PWH). The sessions will provide personalized feedback on alcohol use; a description of adverse effects of alcohol and its role in STI acquisition; a review of reasons to cut down or quit; risky situations, and how to handle them; and optional goal setting. Alcohol-related content of sessions will include reviewing drinking patterns, harmful effects of drinking, and alcohol use behavior change strategies. HIV prevention and treatment content of session will include strategies for increasing HIV care engagement, including ART initiation and adherence and PrEP use for those at risk for HIV. Each session will use cognitive problem solving, skills building, and goal setting to facilitate knowledge, motivation, and behavior to reduce heavy drinking
  Interventions: Behavioral: Treat4All; Behavioral: Standard of care (control arm)
- Standard of care (control arm) (Active Comparator): Participants in the control arm will receive usual care (UC). This includes sexual risk reduction counseling that integrates messaging on reducing alcohol use prior to sex and the recommendation to abstain from alcohol while on ART. Participants in this arm will continue to receive all STI or HIV-related services.
  Interventions: Behavioral: Standard of care (control arm)

INTERVENTIONS:
Behavioral: Treat4All — An alcohol reduction evidence-based intervention integrated with HIV status-neutral counseling
  Arms: Treat4All
Behavioral: Standard of care (control arm) — Sexual risk reduction counseling

SUMMARY:
Purpose: To evaluate short-term efficacy and implementation of Treat4All, an alcohol reduction evidence-based intervention, for decreasing heavy drinking and optimizing HIV outcomes (viral suppression among People with HIV (PWH); Pre-exposure prophylaxis (PrEP) use among those at high risk of HIV)

Participants: Approximately 160 participants aged 18 years or older will be enrolled into this study.

Eligible participants will be recruited from two groups of individuals:

Persons at risk of HIV: Individuals receiving (STI) care who report recent heavy drinking (n=80) and no recent use of PrEP. Persons with HIV: Individuals with HIV who report recent heavy drinking and either a history of unsuppressed viral load or recent suboptimal adherence to ART (n=80).

Procedures (methods): Pilot two-arm randomized controlled trial (1:1; Treat4All Intervention vs Usual Care)

DETAILED DESCRIPTION:
Study Arms

Intervention arm (Treat4All): A total of 80 participants will be randomly allocated to Treat4All. The intervention will be implemented over 3 weeks. Actual session content of Treat4All will vary as a function of an individual's particular issues and HIV status. The intervention will be flexible to allow for discussion of the intersection of alcohol, HIV prevention and treatment, and sexual risk to emerge naturally within the context of the sessions. All sessions will be audiotaped, and a random subsample of 10% will be reviewed to ensure intervention fidelity to core intervention components.

Treat4All will be based on Fleming's Project TrEAT, culturally adapted to the Malawi context, and enhanced to include content on HIV prevention and treatment activities (PrEP use for those at risk for HIV; ART adherence and viral suppression for PWH). The sessions will provide personalized feedback on alcohol use; a description of adverse effects of alcohol and its role in STI acquisition; a review of reasons to cut down or quit; risky situations, and how to handle them; and optional goal setting. Alcohol-related content of sessions will include reviewing drinking patterns, harmful effects of drinking, and alcohol use behavior change strategies. HIV prevention and treatment content of session will include strategies for increasing HIV care engagement, including ART initiation and adherence and PrEP use for those at risk for HIV. Each session will use cognitive problem solving, skills building, and goal setting to facilitate knowledge, motivation, and behavior to reduce heavy drinking and increase engagement in HIV prevention and treatment, including ART adherence and viral suppression among PWH and PrEP use among people at risk for HIV.

Treat4All will consist of three individual in-person weekly sessions, typically 30 minutes each, delivered by a trained counselor. Participants will have 12 weeks after randomization to complete intervention sessions.

Usual care (UC): A total of 80 participants will be randomly allocated to UC. UC includes sexual risk reduction counseling that integrates messaging on reducing alcohol use prior to sex and the recommendation to abstain from alcohol while on ART. This arm will include baseline alcohol and sexual risk assessments, which can itself have an effect on behavior change. By comparing Treat4All to UC, investigators will be able to isolate effects specific to the intervention technique, independent of baseline assessment. Participants in this arm will continue to receive all STI or HIV-related services.

Counseling and linkage to HIV care: All participants, regardless of arm, will receive counseling by a trained HIV counselor. Condoms will be available in each clinic setting. All PWH will be referred to a Lighthouse Trust HIV clinic.

Piloting survey: Investigators will pilot the baseline survey and administration procedures with up to 40 people with similar characteristics to our target population (n=20 PWH; n=20 people at risk for HIV). The pilot will be assessed for survey length and checked for response distribution, item comprehension, and data collection procedures.

Quantitative Assessments: Quantitative assessments will occur at baseline, 3, and 6 months for all participants. All questionnaires will be administered through face-to-face interviews in a private room at the project facility with trained interviewers. Participants who appear influenced by alcohol (assessed by the counselor) or otherwise not lucid will be asked to return for an interview the next day. Study staff will encourage these participants not to drive a motorbike or car from the study site in that state.

Laboratory assessments: HIV viral load, STI testing and dried blood spot collection for alcohol testing will occur at baseline and 6 months.

Screening: Study interviewers will introduce the project to STI clinic patients and, among those who are interested and are 18 years of age or older, interviewers will administer an eligibility written consent to participate in the eligibility screening questionnaire among those who consent.

Enrollment and baseline:

Among those who are eligible for enrollment:

1. Enrollment eligibility will be confirmed using the eligibility screening questionnaire.
2. Enrollment written informed consent will be conducted. Specifically, interviewers will describe the RCT study objectives, procedures, risks and benefits to the eligible participants, and answer any questions. Interviewers will administer the enrollment written informed consent for the client to enroll in the RCT. Once written informed consent is obtained, the participant will be enrolled into the study.
3. Interviewers will collect locator information from the enrolled participant.
4. Interviewers will administer baseline questionnaire
5. Trained laboratory staff will then collect baseline laboratory specimens, including blood and urine, from the enrolled participant.

5. Randomization to Treat4All or usual care

Baseline questionnaire: A quantitative assessment will be performed prior to arm allocation with RCT participants by trained field staff and completed safely and in a confidential place. The survey will be administered to gather information on alcohol use, readiness to change alcohol use, alcohol coping skills, sociodemographic, social desirability, sexual risk, HIV testing history, PrEP use history, PrEP knowledge and willingness, ART initiation, and self-reported ART adherence using the AIDS Clinical Trials Group (ACTG) adherence questionnaire.

Follow-up questionnaires: At months 3 and 6 participants will receive a quantitative follow-up survey that will gather information on: alcohol use, HIV testing history, health status, quality of life, social desirability, readiness to change alcohol use, social support, depression, HIV-related stigma, sexual risk behaviors, PrEP knowledge and willingness, PrEP initiation, and ART initiation and adherence. The research staff will administer all surveys in Chichewa on tablets.

CLINICAL AND LABORATORY EVALUATIONS

Viral load testing: PWH who participant in the RCT (n=80) will have their HIV viral load tested via blood test at baseline and 6 months. Approximately 7.5 milliliters of blood will be drawn for viral load testing. Blood samples will be discarded after viral load testing. Blood samples will be labeled with patient's study ID. The blood draw will take place in a clinic room at the study site and will be conducted by trained clinical staff. HIV-1 RNA level testing will be performed on blood samples at the UNC Project Malawi laboratory according to standard protocols.

Alcohol biomarker: At baseline and month 6, dried blood spots (DBS) will be collected for phosphatidylethanol (PeTH) testing to detect any alcohol use during the 3 weeks before the study visit. Samples will then be kept in drying boxing with a humidity indicator card to monitor moisture levels until they are brought to the laboratory. Samples will be taken to the local laboratory for storage and shipment processing. DBS samples will be sent to the United States for PeTH testing.

STI testing: At baseline and month 6, samples will be collected from all participants with consent and tested for the presence of chlamydia, gonorrhea, and syphilis. Investigators will use the Xpert CT/NG assay, which can be performed on the GeneXpert platform (Cepheid) and is a qualitative, in vitro real-time PCR test for automated detection and differentiation of genomic DNA from chlamydia and/or gonorrhea. Syphilis will be ascertained using a rapid syphilis test, such as the Alere Determine™ Syphilis TP test (Alere Ltd., United Kingdom; sensitivity: 100.0%; specificity: 100.0%).

HIV testing: At month 6, all participants who tested HIV-negative at baseline will be tested for HIV following Malawian National HIV Testing and Counseling guidelines, which indicate serial HIV-antibody rapid tests, such as Determine HIV-1/2 and Uni-Gold rapid HIV-antibody.

Randomization and concealment:

Investigators will complete enrollment and baseline data collection before the assignment of individuals to study arms. Participants will receive the random assignment through prepared envelopes to Treat4All or UC at a ratio of 1:1. Masking of participants and intervention counselors to study arm.

Follow-up questionnaires: At months 3 and 6 participants will receive a quantitative follow-up survey that will gather information on: alcohol use, HIV testing history, health status, quality of life, social desirability, readiness to change alcohol use, social support, depression, HIV-related stigma, sexual risk behaviors, PrEP knowledge and willingness, PrEP initiation, and ART initiation and adherence. The research staff will administer all surveys in Chichewa on tablets.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18 years or older.
* Receiving care at Bwaila STI clinic.
* Report recent heavy drinking (greater than or equal to 4 drinks a day in the past 30 days for men and greater than or equal to 3 drinks a day in the past 30 days for women
* Willing to receive an HIV test at study enrollment, if not previously diagnosed Report not taking ART, recent suboptimal adherence to ART, or recent history of unsuppressed HIV viral load [for PWH] or no recent oral PrEP use (self-reported taking no PrEP pills in past 7 days) [for those at risk of HIV]
* Plan to reside in the Lilongwe area for at least 6 months.
* Not participating in other HIV or alcohol programs
* Ability and willingness of participant to provide informed consent.
* Willingness to provide contact/locator information to be contacted for follow up study activities.

Exclusion Criteria:

* Unable to participate in study activities due to psychological disturbance, cognitive impairment, or threatening behavior
* Pregnant or breastfeeding
* At risk of experiencing alcohol-related withdrawal symptoms
* Acute physical or mental illness, including suicidal thoughts or behaviors
* Participating in in other HIV or alcohol programs
* Active drug dependence that would interfere with adherence to study requirements.
* History of using injectible PrEP
* Any other condition that in the opinion of the study investigator would compromise the safety of the study participant or study staff or would prevent proper conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of heavy drinking days | 6 months after study enrollment
  Proportion of heavy drinking days at month 6 will defined as the proportion of days of heavy drinking (≥4 drinks a day for men and ≥3 drinks a day for women) in the past 21 days. Investigators will collect detailed information on alcohol use through the Alcohol Timeline Follow back (TLFB) to obtain the number of heavy drinking days, percent days abstinent, drinks per drinking day, and measure changes in drinking over time.
Engagement in HIV prevention or treatment | 6 months after study enrollment
  Our co-primary outcome of successful engagement in HIV prevention or treatment will be defined with parallel behaviors across HIV status: PrEP use for people at risk of HIV and viral suppression for PWH. PrEP use will be defined as self-report of >1 pill in the past seven days at month 6. Viral suppression will be defined as an undetectable viral load (<40 copies/mL) at month 6.

SECONDARY OUTCOMES:
STI prevalence | 6 months after study enrollment
  Prevalence of biologically-confirmed STIs (chlamydia, gonorrhea, or syphilis)
ART adherence (among PWH) | ART adherence will be assessed among PWH 6 months after study enrollment
  Self-reported recent ART adherence
HIV incidence | HIV incidence will be assessed 6 months after study enrollment among among participants who tested HIV-negative at study enrollment
  Prevalence of biologically confirmed HIV will be assessed among participants who tested HIV-negative at study enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Parcesepe, PhD, MPH, MSW, Principal Investigator — University of North Carolina, Chapel Hill; Kathryn Lancaster, PhD, Principal Investigator — Wake Forest
Locations (1):
- Bwaila Hospital, Lilongwe, Malawi

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, ICF
Time Frame: beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/ sharing agreement with UNC.

REFERENCES:
- [Derived] Lancaster KE, Bula AK, Matoga MM, Hosseinipour MC, Hoffman IF, Grullon JA, Umar E, Msolola J, Magidson JF, Bonumwezi JL, Hahn JA, Parcesepe AM. Testing a systematically braided alcohol reduction and HIV status neutral intervention among people receiving STI care in Malawi: study protocol for a pilot hybrid type 1 effectiveness-implementation randomized controlled trial. Front Public Health. 2025 Apr 30;13:1572288. doi: 10.3389/fpubh.2025.1572288. eCollection 2025. PMID 40371302